CLINICAL TRIAL: NCT02481973
Title: The Effect of Individualised Homoeopathic Treatment Using the Grant Bentley Method in Premenstrual Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MoniqueChavannes200570791
Record Dates: First submitted 2015-06-04; First posted 2015-06-25 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Premenstrual Syndrome
Keywords: PMS; Homoeopathy; Grant Bentley Method
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individualised Homoeopathic Remedy (Experimental): Each participant is to receive an individualised homoeopathic remedy, prescribed according to their characteristic symptoms and confirmed my their miasmatic facial features. Although different individualised remedies may be dispensed, each remedy will be homoeopathic and prepared in accordance with the German Homoeopathic Pharmacopoeia. Each prescription will be in a potency of 30CH which will be taken once daily, according to the GBM. Sucrose pillules will used as the vehicle for each remedy.
  Interventions: Other: Individualised Homoeopathic Remedy

INTERVENTIONS:
Other: Individualised Homoeopathic Remedy — Each participant is to receive an individualised homoeopathic remedy prescribed according to their characteristic symptoms.

SUMMARY:
Premenstrual syndrome (PMS) is related to the changes in the levels of hormones predominately progesterone, oestrogen and prolactin, during the luteal phase of the menstrual cycle. Both physical and psychological symptoms may occur from at least day 14 of the menstruation cycle and cease by day 4 of menstruation. The symptoms may interfere with a female's daily activities and have a negative impact well-being. There are a number of conventional pharmacological drugs which are used in the treatment or alleviation of the symptoms of PMS, however the drugs may have side effects and may negatively interact with other medications. Research has shown that homoeopathy is beneficial in relieving or decreasing the severity of PMS, however finding the individualised homoeopathic remedy can be difficult. Grant Bentley developed a system that helps find the most suitable remedy for each individual case. The Grant Bentley Method (GBM) uses homoeopathic case taking, photographs of the facial features and repertorisation to determine the dominant miasmatic group of the patient. This aids in the selection of specific homoeopathic remedy. There has been no research to show the effect of the GBM on PMS.

This study aims to determine the effect of individualised homoeopathic treatment using the GBM, on females with PMS by using case studies and a daily self-grading PMS chart.

DETAILED DESCRIPTION:
The study is of an embedded mixed method design using the PMS chart and case studies and will take place over 12 weeks at the University of Johannesburg (UJ) Health Centre. Using purposive sampling, 10 female participants between the ages of 18 to 40 years will be recruited by means of advertisements at the Homoeopathic Health Centre, campus gym and female residences on the Doornfontein campus of the University of Johannesburg, as well as various health shops, practices and gyms in the Auckland Park and Killarney areas, with the relevant permission granted.

Each potential participant will be required to complete a screening questionnaire in order to establish whether they are an appropriate candidate for this study. Once this is confirmed, the researcher will explain the study to each participant. The participants will be required to read the participant information form and sign the consent and medical photograph consent forms. Participants will be informed that their photographs will be used for facial analysis to assist in finding the most accurate remedy and will not be published. Each participant's facial features will be hand-drawn by the researcher in order to aid participant confidentiality.

Each participant will undergo a full homoeopathic consultation which will focus on her PMS symptoms. In addition, 9 photos of their facial features will be taken with a digital camera (Panasonic DMC-FZ5) for classification of their dominant miasmatic group. Thereafter, a physical examination including vital signs and an abdominal and/or breast examination (if indicated) will be conducted.

After the consultation, the participant will be asked to record their daily PMS symptoms, for a period of 1 month, on the PMS chart (provided to them by the researcher) at home. The first month will act as a baseline measurement as no treatment will be prescribed. Additionally, the researcher will analyse and repertorise the participant's case in this period. The participant will be grouped into their dominant miasmatic group and the corresponding remedy will be selected, according to the principles of homoeopathy and GBM of prescribing, for use in the following consultation. Remedy selections will be supervised by a registered homoeopath.

The follow-up consultations will be conducted at weeks 4, 8 and 12, wherein participants will hand in their completed PMS charts and undergo any relevant physical examinations. The participant will then receive their individualised remedy, as determined by the researcher, along with an explanation as to how to store and take the remedy. They will additionally receive another PMS chart to complete over the following 4 weeks. Photographs may be retaken to re-analysed the case if necessary as to ensure the correct selection of the remedy using the GBM during the study.

Should the participant want further treatment at the completion of the study, they will be appropriately referred to a registered homoeopath or to the UJ Homoeopathic Health Centre.

A positive result of this research would indicate the viability of the GBM as a useful tool to aid in the individualised homoeopathic treatment and therefore aid in successful prescribing in the treatment of PMS. Additionally, a positive result would indicate homoeopathy as a potential treatment for PMS.

ELIGIBILITY:
Inclusion Criteria:

* Females (aged 18-40) suffering from at least one PMS symptom from both of the following physical and psychological symptoms, for at least 3 consecutive menstrual cycles:

  * Physical symptoms: headache, breast tenderness, abdominal bloating, food cravings and swelling of extremities
  * Psychological symptoms: depression, anxiety, irritability, social withdrawal and memory changes;
* symptoms that are present from at least day 14 (2 weeks before menstruation) of the menstrual cycle, are relieved by day 4 of menstruation, and do not reoccur until after day 13 of the menstrual cycle; and
* if currently on the OCP, they must be using the same brand of medication for 3 consecutive months.

Exclusion Criteria:

* Females on any kind of chronic medication that may interfere with PMS symptoms such as medication for hyperthyroidism, hypothyroidism, diabetes mellitus and psychiatric disorders;
* are suffering from dysphoric disorder (a severe form of premenstrual syndrome);
* are on hormonal treatment (except OCP);
* have been pre-diagnosed with any anxiety or depression disorders; and/or
* have irregular menses.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
PMS symptom severity as measured by the PMS chart | 12 weeks
  The PMS chart will be conducted daily by each participant for 12 weeks.

SECONDARY OUTCOMES:
Changes in symptom severity as evaluated by researcher case notes | Every 4 weeks for 12 weeks
  Case notes will be taken every 4 weeks in each consultation and will be used to collect qualitative data.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Patel, M.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No